CLINICAL TRIAL: NCT02777684
Title: Motivators and Barriers to Physical Activity in Knee Osteoarthritis Patients: a Qualitative Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Innovatherm (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-0264
Record Dates: First submitted 2016-05-02; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Knee Osteoarthritis
Keywords: Physical activity; Knee osteoarthritis; Non pharmacological treatment; Qualitative study
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- knee osteoarthritis
  Interventions: Other: Qualitative study

INTERVENTIONS:
Other: Qualitative study

SUMMARY:
This study sought to better identify the motivators and barriers to osteoarthritic patients practising regular physical activity. This is a crucial step towards enabling each health professional to adapt their therapy recommendations, while taking into account the patient's overall lifestyle.

DETAILED DESCRIPTION:
The qualitative research design is well-suited to this type of issue. This choice was justified by need to investigate and understand the actions from the participants' point of view. This exploratory method, conducted in the form of individual interviews and focus groups, enabled us to document the personal experiences, practices, and personal history of each individual

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee osteoarthritis

Exclusion Criteria:

-

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Motivators and barriers to physical activity in knee osteoarthritis patients activity | During the spa treatment of 18 days
  Exploratory method, conducted in the form of individual interviews and focus groups enabled us to document the personal experiences, practices, and personal history of each individual (qualitative method)

SECONDARY OUTCOMES:
Definition of physical activity with qualitative method | During the spa treatment of 18 days
Differences between physical activity and sport with qualitative method | During the spa treatment of 18 days
Functional status as assessed by WOMAC | During the spa treatment of 18 days
Level of physical activity with IPAQ short form | During the spa treatment of 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France